CLINICAL TRIAL: NCT03596086
Title: Phase I-II Study Evaluating HSV-tk + Valacyclovir Gene Therapy Combination with Radiotherapy and Chemotherapy for Recurrent Glioblastoma Multiforme
Brief Title: HSV-tk + Valacyclovir + SBRT + Chemotherapy for Recurrent GBM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Baskin MD (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, David Baskin MD, Houston Methodist Neurosurgeon and Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016414
Record Dates: First submitted 2018-03-20; First posted 2018-07-23 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma Multiforme; Astrocytoma, Grade III
Keywords: GBM; glioblastoma; Astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — Genetic Therapy; Genetic Engineering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADV/HSV-tk (gene therapy) (Experimental): The gene therapy investigational product, HSV-tk will be injected during the surgery. Within 24 hours valacyclovir will be given for 14 days. Radiotherapy will be administered over 10 sessions (over 2 weeks) starting within 9 days of surgery. Standard of care/routine chemotherapy will be started concurrent or after completion of the radiotherapy dependent on patient status based on best clinical judgment.
  Patient can receive second treatment of HSV-tk after 6 months
  Interventions: Drug: ADV/HSV-tk (gene therapy)

INTERVENTIONS:
Drug: ADV/HSV-tk (gene therapy) — The investigational adenovirus gene therapy injected at tumor site followed by valacyclovir, radiotherapy, and chemotherapy
  Other Names: gene transfer, gene therapy; HSV-tk

SUMMARY:
Study to assess the safety and efficacy of HSV-tk (gene therapy), valacyclovir, radiotherapy and chemotherapy in recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
This is a prospective phase I-II study to assess the efficacy and toxicity of HSV-tk + valacyclovir gene therapy in combination with radiotherapy in recurrent glioblastoma multiforme or anaplastic astrocytoma. This study is comprised of patients who have failed standard of care treatment (maximal safe resection followed by chemoradiation).

Clinical response will be evaluated by neurological evaluation, neuropsychological testing, and imaging studies as well as by histological examination wherever a re-operation is clinically indicated. Blood samples will be taken for systemic immunological response, blood counts and liver functions tests. Toxicity will be graded by the Common Terminology Criteria for Adverse Events (CTCAE) and Radiation Therapy Oncology Group (RTOG) neuro-toxicity scores. Patients will also be followed to assess median time to progression and median survival.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have biopsy proven recurrent anaplastic astrocytoma or glioblastoma multiforme without evidence of multifocal tumor or brainstem involvement. Multifocal disease does not exist if enhancing areas are connected by abnormal T2 FLAIR on the MRI scan.
* Radiographic evidence of recurrence/progression by iRANO criteria
* ≥ 3 weeks since any major surgery, completion of RT, or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy).
* Life expectancy ≥ 12 weeks.
* Patient can receive second treatment of HSV-tk after 6 months
* Patients should have the following characteristics: recurrent glioblastoma or AA demonstrated by biopsy or imaging study, ECOG performance status of 0-1, has had prior surgery and radiotherapy /chemotherapy for the glioblastoma.
* Patients with leptomeningeal disease may be considered for enrollment into the study.
* No evidence of other active malignancy (except squamous or basal cell skin cancers).
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks of the study by the investigator (or his/her designee) with the aid of written information.
* Willing to provide biopsies as required by the study.
* WOCBP must have a negative serum pregnancy test within 7 days prior to the administration of the first study treatment. Women must not be lactating.
* WOCBP and men must practice an effective method of birth control
* Patients must have adequate baseline organ function as assessed by the following laboratory values before initiating the protocol:

  * serum creatinine < 1.5 mg/dL
  * T. bilirubin < 2.5 mg/dL, ALT, AST, GGT and AP < 2 x normal
  * Platelet count. > 100,000/ml , ANC> 1500/ml , Hgb> 10 gm/dL
  * Normal partial thromboplastin time (PTT) and Pro-Thrombin Time (PT)
* Non English speaking patients can participate in this study

Exclusion Criteria

* Prior treatment with immunomodulatory therapy, immunotherapy, and/or gene vector therapy in the past 3 months.
* Any cytotoxic chemotherapy, RT, or immunotherapy or any investigational drug for this brain tumor within 3 weeks of study treatment start.
* Evidence of multifocal disease, brainstem involvement
* Patients on immunosuppressive drugs (other than steroids for brain edema).
* In patients with leptomeningeal disease, no evidence of diffuse disease or spread to the spine.
* In patients with leptomeningeal disease, no bulky leptomeningeal metastases with potential to obstruct CSF flow will not be enrolled.
* Liver disease, such as cirrhosis or active/chronic hepatitis B or C.
* History of or current alcohol misuse/abuse within the past 12 months.
* Known or suspected allergy or hypersensitivity to any component of the proposed regimen (gene vector-HSV-tk, Valacyclovir).
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications (Valacyclovir).
* No active malignancy except for non-melanoma skin cancer or in situ cervical cancer or treated cancer from which the patient has been continuously disease free for more than 5 years.
* Pregnant or breastfeeding women or women/men able to conceive and unwilling to practice an effective method of birth control. WOCBP must have a negative serum pregnancy test within 7 days prior to the administration of the first study treatment.
* Presence of active or suspected acute or chronic uncontrolled infection or history of immunocompromise, including a positive HIV test result.
* Patients < 18 years of age
* Unwilling or unable to comply with the study protocol.
* The presence of active CNS toxoplasmosis infection or Progressive Multifocal Leukoencephalopathy demonstrated on CT or MRI imaging.
* The presence of active untreated cellulitis or untreated wound infections. Treated and resolving cellulitis and infections are not an exclusion criteria.
* Active IV drug abuse or severe opioid abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival in months from Study drug administration (Day 0) | Up to 60 months as measured in months.
  The overall survival in months of recurrent GBM patients drug administration up to five years

SECONDARY OUTCOMES:
Progression Free Survival assessments will be done every 6-8 weeks for 1st year thereafter every 12-14 weeks until disease progression or death | Up to 60 months as measured in months
  Patients will have MRI or CT every 6-8 weeks for the first year post surgery. Thereafter patient will have MRI or CT every 12-14 weeks until completion of the protocol study specific treatment. Progression free survival will be assessed by RANO response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: David S Baskin, MD, Principal Investigator — Houston Methodist Neurological Institute
Locations (1):
- Houston Methodist Neurological Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined